CLINICAL TRIAL: NCT02794623
Title: Evaluation of Tinnitus Suppression for Cochlear Implant Recipients
Brief Title: Tinnitus Suppression for Cochlear Implant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Royal Victoria Eye and Ear Hospital (Other Government); Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC 5583
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Tinnitus
Keywords: cochlear implants; hearing loss
MeSH Terms: conditions — Tinnitus; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear Implant Recipients (Experimental)
  Interventions: Device: Tinnitus masking

INTERVENTIONS:
Device: Tinnitus masking — Tinnitus masking via CI system

SUMMARY:
Tinnitus is the perception of sound in the absence of an external sound. Prevalence in the general population is 10 to 15%, with tinnitus severely impacting quality of life in 1-2 percent of the population. Tinnitus therapy is based on counselling, cognitive and behavioural therapies in combination with sound therapies which mostly rely on masking.

For cochlear implant candidates, the ability to use hearing aids and maskers is limited by the degree of their hearing loss. Reports of tinnitus prevalence in this group range from 67 to 100% with a mean of 80%.

In cochlear implant (CI) recipients, tinnitus suppression primarily occurs during active use of the cochlear implant system. In some CI recipients residual inhibition of tinnitus occurs when the implant is switched off. While the benefits of CI implantation on tinnitus are well documented, there is a group of recipients where tinnitus remains a concern in the implanted ear post-operatively.

The primary aim of this study is to investigate the benefits of using tinnitus masking via a CI sound processor that optimises tinnitus suppression with minimal annoyance to the user. Furthermore a questionnaire will be employed to capture the prevalence, degree and nature of tinnitus in recipients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Freedom or CI500 series implant
3. At least 3 months experience with the cochlear implant
4. Native speaker in the language used to assess speech perception performance
5. Willingness to participate in and to comply with all requirements of the protocol
6. Self-reported tinnitus in the implanted ear
7. Reside local to investigational site

Exclusion Criteria:

1. Signs of retrocochlear or central origin to hearing impairment as confirmed by medical examination and test including MRI
2. Additional handicaps that would prevent participations in evaluations
3. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10-18 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Tinnitus Severity Questionnaire | Testing over 6 months
  Tinnitus severity questionnaire using Visual Analog Scale
Word recognition scores in quiet | Testing over 6 months
  Monosyllabic word scores in quiet
Speech recognition scores in noise | Testing over 6 months
  Sentence recognition scores in noise

SECONDARY OUTCOMES:
Degree of handicap as a result of tinnitus | Testing over 6 months
  Tinnitus Handicap Questionnaire used to capture degree of overall handicap as a result of tinnitus

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No